CLINICAL TRIAL: NCT01177202
Title: A Phase I Dose-Escalation Study to Investigate the Safety and Immunogenicity of the Fusion Protein Recombinant Influenza A (HAC1) Vaccine Derived From Influenza A/California/04/09 (H1N1) in Healthy Adults
Brief Title: Study of the Safety and Immunogenicity of H1N1 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fraunhofer, Center for Molecular Biotechnology (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: WRAIR 1758
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: H1N1 Flu
Keywords: HAC1, H1N1
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group A (Experimental): HAC1 Dose = 15ug; Alum Dose = 0
  Interventions: Biological: HAC1 Vaccine
- Group B (Experimental): HAC1 Dose = 15ug; Alum Dose = 0.75mg
  Interventions: Biological: HAC1 Vaccine
- Group C (Experimental): HAC1 Dose = 45ug; Alum Dose = 0
  Interventions: Biological: HAC1 Vaccine
- Group D (Experimental): HAC1 Dose = 45ug; Alum Dose = 0.75mg
  Interventions: Biological: HAC1 Vaccine
- Group E (Experimental): HAC1 Dose = 90ug; Alum Dose = 0
  Interventions: Biological: HAC1 Vaccine
- Group F (Experimental): HAC1 Dose = 90ug; Alum Dose = 0.75mg
  Interventions: Biological: HAC1 Vaccine
- Group G (Placebo Comparator): Saline
  Interventions: Biological: HAC1 Vaccine
- Group H (Active Comparator): H1N1
  Interventions: Biological: HAC1 Vaccine

INTERVENTIONS:
Biological: HAC1 Vaccine — Subjects will come to the Clinical Trials Center up to 7 days prior to each vaccine dose to have blood drawn for research assays. The first dose of vaccine will be given on Day 0 and the second dose will be given 21 days later (± 3 days). Dose escalation will be staggered by at least 7 days as shown in Figure 1. Subjects from Groups G and H will be vaccinated with each of the other 6 groups. Two subjects from group A will be immunized on study day -1. The immunizations will be performed one hour apart with close monitoring. The remaining eight subjects from Group A will be immunized on study day 0. All subsequent immunizations for each group will occur on the same day. The principal investigator and the medical monitor will review all adverse events and make a determination on whether it is safe to proceed to the next higher dosage group. The control and reference vaccine groups can be vaccinated starting anytime after screening.

SUMMARY:
The Purpose Of This Study Is To Assess The Safety, Immunogenicity, And Tolerability Of A H1N1 Vaccine In Healthy Adults

DETAILED DESCRIPTION:
This is a single center, placebo-controlled, single blinded dose escalation study to preliminarily assess the safety, reactogenicity, and immunogenicity of different HAC1 vaccine formulations. This study will assess a novel HAC1 vaccine, which is plant derived. This vaccine will be compared to Placebo of normal (0.9%) saline, and reference vaccine consisting of an approved monovalent vaccine containing an A/California (H1N1)-like strain.

Subjects will receive 2 intramuscular injections of the experimental vaccine, placebo, or reference vaccine on Study Days 0 and 21

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 50 years inclusive
* Able to give written informed consent to participate
* Score of at least 80% correct on a 10 question multiple-choice quiz (2 attempts)
* Healthy, as determined by medical history, physical examination, weight, vital signs, and clinical safety laboratory examinations at baseline
* Females must fulfill one of the following criteria: At least one year post-menopausal; Surgically sterile or have a surgically sterile partner; Willing to abstain from sexual intercourse; Willing to use a reliable form of contraception approved by the investigator (e.g., oral, implantable, transdermal or injectable contraceptives, intrauterine device (IUD), female condom, diaphragm with spermicide, cervical cap, or male condoms) for 30 days prior to first vaccination through 3 months after second vaccination
* Women of childbearing potential must have a negative urine pregnancy test within 24 hours preceding receipt of each dose
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits and to be contacted by telephone throughout the follow-up period

Exclusion Criteria:

* Prior receipt of 2010-2011 seasonal influenza vaccine containing A/California/04/09-like virus
* Screening H1N1 titer of > 1:40
* Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical or surgical treatment or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening
* Presence of any medical condition that may be associated with impaired immune responsiveness, including diabetes mellitus
* Cancer, or treatment for cancer, within the previous 3 years, excluding basal cell carcinoma or squamous cell carcinoma
* Presently receiving or history of receiving, during the preceding 3-month period, any medications or other treatments that may adversely affect the immune system: This includes allergy injections, immune globulin, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable); Inhaled and topical corticosteroids will be allowed
* Receipt of blood or blood products 8 weeks prior to vaccination or planned administration during the study period
* Donation of blood or blood products within 8 weeks prior to vaccination or at any time during the study
* Receipt or planned administration of a nonstudy vaccine within 30 days prior to vaccination; Immunization on an emergency basis with Tetanus Toxoids Adsorbed for adult use (Td or Tdap) vaccine up to 8 days before or at least 8 days after a dose of study vaccine will be allowed
* History of anaphylactic type reaction to injected vaccines
* Receipt of any investigational product or nonregistered drug within the 30 days prior to vaccination or currently enrolled in any investigational drug study or intends to enroll in such a study within the ensuing study period
* History of drug or chemical abuse in the year before the study
* Positive serology for HIV-1 or HIV-2, or HBsAg or HCV antibodies
* Unwilling to allow storage of specimens for future use
* Acute disease within 72 hours prior to vaccination: Acute disease is defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical examination) with or without fever (>38ºC />100.4ºF), or an oral temperature of >38ºC orally; Study vaccine can be administered to persons with a minor illness.
* Any condition that, in the opinion of the investigator, might interfere with interpretation of data supporting the primary study objectives

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess the safety, reactogenicity, and tolerability of the HAC1 vaccine formulations. | Six Months
  The primary objective of this study is to assess the safety, reactogenicity, and tolerability of the HAC1 vaccine formulations delivered intramuscularly at doses of 15 μg, 45 μg or 90 µg (unadjuvanted or adjuvanted) in healthy adults 18 - 50 years of age.

SECONDARY OUTCOMES:
To assess and compare the immunogenicity to 2 injections of the 6 HAC1 vaccine formulations. | Six Months
  The secondary objective is to assess and compare the immunogenicity to 2 injections of the 6 HAC1 vaccine formulations using existing research assays and by measuring hemagglutination inhibition (HAI) titers.

CONTACTS AND LOCATIONS:
Overall Officials: James F Cummings, MD, LTC(P), MC, USA, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research (WRAIR), Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cummings JF, Guerrero ML, Moon JE, Waterman P, Nielsen RK, Jefferson S, Gross FL, Hancock K, Katz JM, Yusibov V; Fraunhofer USA Center for Molecular Biotechnology Study Group. Safety and immunogenicity of a plant-produced recombinant monomer hemagglutinin-based influenza vaccine derived from influenza A (H1N1)pdm09 virus: a Phase 1 dose-escalation study in healthy adults. Vaccine. 2014 Apr 17;32(19):2251-9. doi: 10.1016/j.vaccine.2013.10.017. Epub 2013 Oct 12. PMID 24126211